CLINICAL TRIAL: NCT03886675
Title: Carbon-Dioxide Flushing Versus Saline Flushing in Thoracic Endovascular Aortic Repair to Reduce Neurological Injury: A Pilot Randomised Controlled Trial
Brief Title: Intervention With Cerebral Embolic Protection in TEVAR: Gaseous Protection
Acronym: INTERCEPT:GP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); South Canterbury DHB, New Zealand (Unknown); Baylor Scott and White Health (Other); University Hospital Southampton NHS Foundation Trust (Other); Health New Zealand (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INTERCEPT:GP
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Silent Cerebral Infarction; Neurocognitive Dysfunction; Vascular Brain Injury
Keywords: Stroke; Silent cerebral infarction; Carbon dioxide; Thoracic endovascular aortic repair; TEVAR; DW-MRI; Vascular brain infarction
MeSH Terms: conditions — Stroke; Cognition Disorders; Cerebrovascular Trauma

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to treatment allocation. Assessment of TCD embolic data, DW-MRI scan reporting and neurological and neurocognitive assessment will be carried out by blinded trained assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbon-dioxide (Experimental): Flushing of stent-grafts in TEVAR with carbon-dioxide
  Interventions: Other: CO2 flushing
- Saline (Active Comparator): Flushing of stent-grafts with saline
  Interventions: Other: Saline flushing

INTERVENTIONS:
Other: CO2 flushing — As above
  Arms: carbon-dioxide
Other: Saline flushing — As above
  Arms: Saline

SUMMARY:
Vascular brain infarction (VBI) occurs in 67% of patients undergoing TEVAR. Overt stroke occurs in 13% of these patients and 88% of patients suffer from neurocognitive impairment.

Cerebral air embolisation during the stent-graft deployment phase of TEVAR may be a cause of VBI. Standard treatment to de-air stent-grafts is through the use of a saline flush.

This study aims to investigate whether carbon-dioxide or saline is the better fluid to de-air TEVAR stent-grafts prior to insertion in to the patient and compare VBI rate in the carbon-dioxide group and saline group.

DETAILED DESCRIPTION:
Thoracic endovascular aortic repair (TEVAR) is the re-lining of the thoracic aorta to prevent life threatening haemorrhage and death from rupture. This involves a small cut in the femoral artery in the groin and under imaging guidance, the insertion of wires and a stent into the thoracic aorta.

Prior to insertion into the patient, stents are flushed with saline to remove air and prevent air reaching the brain that can cause a form of brain injury known as vascular brain infarction (VBI). However, our preliminary clinical data suggests that saline flushing is not effective at de-airing stent-grafts used in TEVAR.

Carbon-dioxide has been used extensively in cardiac surgery to displace air from the chest cavity to prevent peri-procedural cerebral air embolisation. We hypothesise that flushing the stent-grafts with carbon-dioxide may be better at removing air from the stent-grafts than saline flush.

Patients undergoing TEVAR will be approached to participate in this study. After written consent is obtained, participants will be randomised to undergo (TEVAR) with carbon dioxide or saline flushing of stent-grafts. Pre-operatively, participants will undergo extensive neurocognitive testing, and a baseline blood test. Intra-operatively, participants will undergo continuous transcranial doppler monitoring (TCD) of the middle cerebral artery (MCA) to look for cerebral air embolisation at stent-graft deployment phase of TEVAR. Blood testing pre-op, immediately post op, and 24 hours post op will be taken to measure for biomarkers of brain injury. Post-operatively, participants will undergo another diffusion-weighted brain MRI within 72 hours post-procedure, stroke and delirium assessment at day 1, 3 and day 7 +/- day of discharge, and at 6-weeks and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All participants suitable for TEVAR with capacity to consent

Exclusion Criteria:

* Participants who lack capacity to consent
* Contraindications to MRI such as pacemaker
* Pregnant participants
* Participants who do not wish to participate
* Participants <18yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-06-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 36 months
  The number of patients recruited into the trial will be collected
Retention | 36 months
  The proportion of patients undergoing follow-up assessments will be collected
Study design for full randomised controlled trial | 36 months
  The proportion of patients who are eligible for the trial will be collected

SECONDARY OUTCOMES:
Number, size and location of new ischaemic lesions on post-operative diffusion-weighted MRI scans | 36 months
  Using DW-MRI at <72 hours post operatively (day 1-7), and also 6 months post operatively, we will assess for new ischaemic lesions
Number of gaseous and solid intra-operative transcranial doppler microembolic signals by phase of TEVAR | Duration of surgery, 36 months collection
  At all London units, transcranial doppler insonation of the middle cerebral artery will be carried out during the procedure, and analysed offline at a later date to evaluate gaseous or solid emboli during TEVAR
Number of participants with stroke or delirium as an inpatient | These will be carried out within 48 hours of patients' return to level 1 care. 36 months collection
  Patients will undergo stroke and delirium assessment.
Serial biomarker blood tests | 36 months
  Blood samples will be taken preoperatively, at the end of the procedure and 24 hours late. These will be analysed for a biomarker of neuroglial injury, S100B
Risk factor assessment | 36 months
  Data such as stent type will be collected.
Neurological assessment, delirium assessment and quality of life testing | Pre-op, first outpatient assessment (approximately 6 weeks), 6 months. 36 months collection
  Patients will undergo a baseline neurocognitive, delirium and quality of life testing. These will be repeated as an outpatient to measure change post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gibbs, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be made to the corresponding author and make on a case by case basis
Supporting Information: Study Protocol, ICF
Time Frame: 10 years
Access Criteria: These will be reviewed on a case by case basis

REFERENCES:
- [Background] Perera AH, Rudarakanchana N, Monzon L, Bicknell CD, Modarai B, Kirmi O, Athanasiou T, Hamady M, Gibbs RG. Cerebral embolization, silent cerebral infarction and neurocognitive decline after thoracic endovascular aortic repair. Br J Surg. 2018 Mar;105(4):366-378. doi: 10.1002/bjs.10718. Epub 2018 Feb 12. PMID 29431856
- [Background] Kahlert P, Eggebrecht H, Janosi RA, Hildebrandt HA, Plicht B, Tsagakis K, Moenninghoff C, Nensa F, Mummel P, Heusch G, Jakob HG, Forsting M, Erbel R, Schlamann M. Silent cerebral ischemia after thoracic endovascular aortic repair: a neuroimaging study. Ann Thorac Surg. 2014 Jul;98(1):53-8. doi: 10.1016/j.athoracsur.2014.03.037. Epub 2014 May 17. PMID 24841546
- [Background] Masada K, Kuratani T, Shimamura K, Kin K, Shijo T, Goto T, Sawa Y. Silent cerebral infarction after thoracic endovascular aortic repair: a magnetic resonance imaging study. Eur J Cardiothorac Surg. 2019 Jun 1;55(6):1071-1078. doi: 10.1093/ejcts/ezy449. PMID 30629169
- [Background] Inci K, Koutouzi G, Chernoray V, Jeppsson A, Nilsson H, Falkenberg M. Air bubbles are released by thoracic endograft deployment: An in vitro experimental study. SAGE Open Med. 2016 Dec 7;4:2050312116682130. doi: 10.1177/2050312116682130. eCollection 2016. PMID 27994872
- [Background] Rohlffs F, Tsilimparis N, Saleptsis V, Diener H, Debus ES, Kolbel T. Air Embolism During TEVAR: Carbon Dioxide Flushing Decreases the Amount of Gas Released from Thoracic Stent-Grafts During Deployment. J Endovasc Ther. 2017 Feb;24(1):84-88. doi: 10.1177/1526602816675621. Epub 2016 Oct 26. PMID 27798380
- [Background] Martens S, Neumann K, Sodemann C, Deschka H, Wimmer-Greinecker G, Moritz A. Carbon dioxide field flooding reduces neurologic impairment after open heart surgery. Ann Thorac Surg. 2008 Feb;85(2):543-7. doi: 10.1016/j.athoracsur.2007.08.047. PMID 18222261
- [Background] Ganguly G, Dixit V, Patrikar S, Venkatraman R, Gorthi SP, Tiwari N. Carbon dioxide insufflation and neurocognitive outcome of open heart surgery. Asian Cardiovasc Thorac Ann. 2015 Sep;23(7):774-80. doi: 10.1177/0218492315583562. Epub 2015 May 4. PMID 25939908
- [Background] Bismuth J, Garami Z, Anaya-Ayala JE, Naoum JJ, El Sayed HF, Peden EK, Lumsden AB, Davies MG. Transcranial Doppler findings during thoracic endovascular aortic repair. J Vasc Surg. 2011 Aug;54(2):364-9. doi: 10.1016/j.jvs.2010.12.063. Epub 2011 Mar 3. PMID 21371850
- [Derived] Crockett S, Hanna L, Singh A, Gunning S, Nicholas R, Bicknell C, Hamady M, Gable D, Sallam M, Modarai B, Abisi S, Lyons O, Gibbs R. Carbon dioxide flushing versus saline flushing of thoracic aortic stents (INTERCEPTevar): protocol for a multicentre pilot randomised controlled trial. BMJ Open. 2023 Apr 27;13(4):e067605. doi: 10.1136/bmjopen-2022-067605. PMID 37105705